CLINICAL TRIAL: NCT00323466
Title: A Study of the Effect on Oro-dental Complications of Intensity Modulated Radiotherapy (IMRT) Versus Conventional Radiotherapy in Patients With Cancer of the Head or Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/164
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cancer: Head or Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT (Experimental)
  Interventions: Procedure: IMRT versus conventional radiotherapy

INTERVENTIONS:
Procedure: IMRT versus conventional radiotherapy — Comparing MRT versus conventional radiotherapy

SUMMARY:
Study to investigate the effect of two types of radiotherapy on saliva: IMRT versus conventional radiotherapy.

In each group, one part will receive normal dental preventive treatment. The other part will use products for treatment of dry mouth (Biotene gamma).

Both anorganic and organic components of the saliva will be studied at different time points, combined with bacterial swabs.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Cancer of head or neck

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Volume of saliva | Before, during (week 4) and after radiation (week 2, 3, 6 and 12)
Quality of saliva | Before, during (week 4) and after radiation (week 2, 3, 6 and 12)
Oral flora | Before, during (week 4) and after radiation (week 2, 3, 6 and 12)

CONTACTS AND LOCATIONS:
Overall Officials: Roeland De Moor, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be